CLINICAL TRIAL: NCT07302789
Title: Clinical Evaluation of the Improvement of Skin Beauty Parameters After Oral Intake of a Collagen Peptides Supplement in Human Volunteers
Brief Title: Clinical Effects of Two Oral Bioactive Collagen Peptides On Skin Properties and Aging Hallmarks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bionos Biotech S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Collagen peptides suppl_2025
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Skin Ageing; Facial Wrinkles - Rough Texture - Hyperpigmentation; Skin Hydration in Healthy Volunteers
Keywords: Collagen peptides; Oral collagen supplement; Skin aging; Facial wrinkles; Skin elasticity; Skin firmness; Skin hydration; Transepidermal water loss (TEWL)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was conducted as a double-blind, parallel-group cosmetic trial. The investigational collagen peptides supplement and the comparator collagen supplement were packaged and labeled as "Product A" and "Product B," so that participants, care providers, investigators, and outcomes assessors were all unaware of group assignment. The treatment code was held by the sponsor/designee and was not broken until completion of data collection and database lock, except in case of a medical emergency requiring individual unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Peptides Supplement (Experimental): 34 healthy women aged 35-65 years with visible wrinkles in the crow's-feet area receive a daily oral collagen peptides supplement for 8 weeks. Participants take one sachet per day while maintaining their usual diet and skincare routines and avoiding new oral supplements or intensive cosmetic procedures.
  Interventions: Other: Dietary Supplement: Collagen Peptides Supplement
- Competitor's Collagen Supplement (Active Comparator): 33 healthy women aged 35-65 years with visible wrinkles in the crow's-feet area receive a daily oral competitor collagen supplement for 8 weeks. Participants take one sachet per day while maintaining their usual diet and skincare routines and avoiding new oral supplements or intensive cosmetic procedures.
  Interventions: Other: Dietary Supplement: Competitor's Collagen Supplement

INTERVENTIONS:
Other: Dietary Supplement: Collagen Peptides Supplement — Participants will be provided with the Collagen peptides supplement and instructed to take one sachet orally once daily for 8 weeks (one 2,500 mg sachet diluted in water or another beverage, preferably in the morning at approximately the same time each day). Efficacy will be evaluated at baseline and at approximately 4 and 8 weeks after the first intake by measuring facial skin elasticity, firmness, and fatigue with a Cutometer®, wrinkle area/depth/volume in the crow's-feet region with VISIA-CR®/PRIMOS® 3D imaging, skin hydration with a Corneometer®, and skin barrier function (transepidermal water loss) on the cheek with a Tewameter®. The product is a pure hydrolyzed bovine collagen peptides powder (2,500 mg per sachet), free of artificial additives/E-numbers and compliant with EU food regulations. All procedures and instrumental measurements take place at Bionos Biotech S.L. facilities.
  Arms: Collagen Peptides Supplement
Other: Dietary Supplement: Competitor's Collagen Supplement — Participants will be provided with the Competitor's collagen supplement and instructed to take one sachet orally once daily for 8 weeks (one 2,500 mg sachet diluted in water or another beverage, preferably in the morning at approximately the same time each day). Efficacy will be evaluated at baseline and at approximately 4 and 8 weeks after the first intake using the same non-invasive methods: Cutometer® (elasticity, firmness, fatigue), VISIA-CR®/PRIMOS® 3D imaging (crow's-feet wrinkle area, depth, and volume), Corneometer® (facial skin hydration), and Tewameter® (transepidermal water loss on the cheek). The product is a pure hydrolyzed bovine collagen peptides powder (2,500 mg per sachet), currently marketed as a collagen supplement and compliant with international food-safety regulations. All procedures and instrumental measurements take place at Bionos Biotech S.L. facilities.
  Arms: Competitor's Collagen Supplement

SUMMARY:
This randomized, controlled clinical trial evaluated whether daily oral intake of a collagen peptides supplement improved age-associated skin beauty parameters in healthy women with visible facial wrinkles. A total of 68 healthy female volunteers between 35 and 65 years of age (both inclusive) with noticeable facial wrinkles were initially enrolled in this randomized, double-blind, parallel-group clinical study. Participants were allocated in a 1:1 ratio to receive either the active control (n = 34) or avvera™ (n = 34). One participant in the active control group withdrew from the study due to personal reasons and was excluded from the final analysis. Consequently, 67 participants completed the study and were included in the efficacy analyses (active control: n = 33; avvera™: n = 34). Participants consumed one 2,500 mg sachet per day, diluted in water or another beverage, while maintaining their usual diet and skincare routines and avoiding other oral supplements or intensive cosmetic procedures for 8 weeks.

The main objectives were to determine whether each collagen supplement, considered independently, (1) improved facial skin elasticity, firmness, and fatigue; (2) reduced wrinkle area, depth, and volume in the crow's-feet region; and (3) enhanced skin hydration and barrier function. At baseline (Day 0) and at weeks 4 and 8, participants attended clinic visits where skin elasticity, firmness, and fatigue were measured with a Cutometer; wrinkles were assessed by VISIA-CR/PRIMOS imaging; skin hydration was measured with a Corneometer; and transepidermal water loss on the cheek was quantified with a Tewameter. The study was designed to assess the efficacy of each product separately, without formal head-to-head comparison between them.

DETAILED DESCRIPTION:
Skin aging is a multifactorial process driven by intrinsic factors (genetic background, hormonal changes, chronological aging) and extrinsic factors such as UV exposure, environment, and lifestyle. Clinically, it is characterized by wrinkles, loss of elasticity and firmness, decreased hydration, and impaired barrier function. Nutraceuticals are increasingly used as complementary strategies to support skin health from within, and hydrolyzed collagen has emerged as a particularly promising ingredient. Collagen peptides derived from bovine hide and processed by enzymatic hydrolysis yield bioactive fragments with good bioavailability and regulatory recognition as safe ingredients for long-term oral intake. However, additional controlled clinical studies were needed to further substantiate their cosmetic benefits on age-related skin parameters.

This double-blind, parallel-group cosmetic clinical study was conducted at Bionos Biotech S.L. (Valencia, Spain) to evaluate the effects of daily oral intake of an Italgel S.p.A. Collagen peptides supplement on facial skin beauty parameters in comparison with a commercially available Competitor's supplement. Sixty-eight healthy female volunteers aged 35-65 years with visible wrinkles in the crow's-feet area were enrolled after meeting predefined inclusion and exclusion criteria and signing written informed consent. Participants were allocated in a 1:1 ratio to receive either the active control (n = 34) or avvera™ (n = 34). One participant in the active control group withdrew from the study due to personal reasons and was excluded from the final analysis. Consequently, 67 participants completed the study and were included in the efficacy analyses (active control: n = 33; avvera™: n = 34). Key exclusions included relevant systemic diseases, abnormal liver or kidney function, heavy alcohol intake, current smoking or recent smoking history, use of certain systemic medications (e.g., oral hormones, steroids, obesity drugs, antidepressants), and conditions judged by the investigator as incompatible with participation. Eligible participants were assigned to receive either the Collagen peptides supplement or the Competitor's supplement (30 women per group) for 8 weeks.

Both investigational products consisted of pure hydrolyzed bovine collagen supplied in sachets containing 2,500 mg of powder. The collagen was manufactured under European food-safety regulations, using enzymatic hydrolysis to obtain small peptides with high absorption and without added artificial ingredients or E-numbers. Products were labeled as "Product A" and "Product B" so that neither volunteers nor investigators knew which product each participant was taking; the identity code was held by the sponsor. Participants were instructed to dissolve one sachet per day in water or another beverage and to ingest it once daily, preferably in the morning at approximately the same time, for a total of 8 consecutive weeks.

Efficacy assessments focused on objective, non-invasive measurements of skin mechanics, wrinkles, hydration, and barrier function. At baseline (Day 0), Week 4, and Week 8, participants attended clinic visits in which facial skin elasticity, firmness, and fatigue were quantified using a Cutometer®; wrinkle area, depth, and volume in the crow's-feet region were analyzed by 3D imaging with VISIA-CR/PRIMOS technology; stratum corneum hydration on the face was measured by Corneometer®; and transepidermal water loss (TEWL) on the cheek was assessed using a Tewameter®. These time points allowed evaluation of changes over time within each treatment group as well as comparison of responses between the Collagen peptides supplement and the Competitor's supplement.

Throughout the study, volunteers were asked to maintain their usual eating habits and basic skincare routines and to avoid starting any new oral supplements (including antioxidants or other "beauty from within" products) that could interfere with interpretation of results. Participants were allowed to continue their regular day and night topical care, but they were instructed not to undergo intensive or invasive cosmetic procedures (such as strong peels, aggressive masks, or similar treatments) during the study. Major changes in personal cosmetic routines or lifestyle that might impact study endpoints were discouraged, and contraceptive methods were to remain stable. Compliance with product use and adherence to study instructions were supported through written guidelines and close contact with the research team.

Safety was monitored throughout the 8-week intervention. Hydrolyzed collagen is widely used in supplements and is generally regarded as safe, and no health risks were anticipated at the doses used. Nevertheless, volunteers were instructed to seek medical attention immediately if they experienced any adverse events, and the attending healthcare professionals could recommend temporary or permanent discontinuation of the product if needed. All adverse events and any serious undesirable events were to be documented and reported to the sponsor and ethics committees according to regulatory timelines, and participants who discontinued were followed until resolution of any study-related effects.

For the analysis, results obtained before and after supplementation were used to determine the effects of oral collagen intake on the different skin parameters. Data were analyzed statistically using an unpaired Student's t-test with a two-sided significance level of 0.05 (95% confidence interval). Based on prior experience of Bionos Biotech S.L. in similar clinical studies, a total sample size of 60 women (30 per group) was considered sufficient to detect differences on the order of approximately 5-10% with 80% power, while acknowledging that exact effect sizes could not be predicted in advance. The study was primarily designed to characterize the efficacy profile of each collagen supplement; any comparative interpretation between products was to be made by the sponsor.

The trial was conducted in accordance with the Declaration of Helsinki, ICH guidelines, and applicable national regulations. The protocol, informed consent document, and study materials were reviewed and approved by the relevant Ethics Committee in Clinical Research and the regional health authority of the Generalitat Valenciana before initiation. All participants provided written informed consent prior to any study procedures. Study data were recorded in source documents and case report forms and then coded to protect participant identity in line with Spanish data protection legislation; the sponsor had access only to anonymized study data. Essential documents, signed consent forms, and accountability records for the investigational products were retained by the investigator in accordance with regulatory requirements and the sponsor's policies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female volunteers.
* Between 35-65 years old (both included).
* With noticeable wrinkles (wrinkles in the crow's feet area).
* Subjects with absence of any infectious disease within the 4 weeks previous to the study.
* Informed of the purpose and the protocol of the study and signed a written informed-consent form.

Exclusion Criteria:

* Diagnosis of any diseases such as cardiovascular disease, chronic kidney disease (CKD), gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease.
* Consume more than the recommended alcohol guidelines i.e. >14 units/week for females (europa.eu).
* Current smoking habit or history of smoking within the past 1 year.
* History of depression, schizophrenia, alcoholism, drug addiction, or mental illness.
* Current or previous intake of contraceptives, female hormones, obesity drugs, absorption inhibitors, antidepressants, or appetite suppressants.
* History of asthma or autoimmune disease Use of oral hormone therapies ie. cortisone or steroids in the 6 months prior to initiation of the study.
* Abnormal liver function or abnormal renal function.
* Blood pressure >140/90 mmHg or hypertension with intake of a diuretic.
* Any condition judged by the investigator to be unsuitable for participation in the study.

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Actual)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Quantification of the change in facial wrinkle parameters (area, length, depth, and volume) in the crow's-feet region from baseline to post-treatment visits using 3D imaging. | Baseline (Day 0) and at approximately Day 28 (~4 weeks) and Day 56 (~8 weeks) of treatment.
  Sixty healthy women (35-65 years) with visible wrinkles in the crow's-feet area will take either a Collagen peptides supplement or a Competitor's collagen supplement once daily for 8 weeks. Facial wrinkles, with emphasis on crow's feet, will be assessed using the Visia-CRP-5 Primos system (Canfield Scientific, USA). Standardized images (clean skin, closed eyes, neutral expression) will be captured at three angles (left 45°, frontal, right 45°) using a stabilization rig. 3D reconstructions will be analyzed to quantify wrinkle area, length, depth, and volume in predefined regions of interest. Changes in these parameters from baseline to post-treatment visits will be calculated within each treatment group. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; products are supplied in individual single-dose sachets and stored according to the manufacturer's instructions.
Quantification of the change in facial skin firmness, elasticity, and fatigue from baseline to post-treatment visits using Cutometer®. | Baseline (Day 0, before product intake) and at approximately Day 28 (~4 weeks) and Day 56 (~8 weeks) of treatment
  Sixty healthy women (35-65 years) with visible wrinkles in the crow's-feet area will take either a Collagen peptides supplement or a Competitor's collagen supplement once daily for 8 weeks (one 2,500 mg sachet diluted in water or another beverage, preferably in the morning at approximately the same time each day). Facial skin mechanical properties will be quantified using a Cutometer® MPA 580 (Courage + Khazaka, Cologne, Germany), which applies controlled negative pressure to the skin and optically records vertical displacement. Firmness (R0), elasticity (R5), and skin fatigue/viscoelastic "tiring" (R3) will be derived from the deformation-recovery curve. Measurements will be taken on the cheek of each volunteer at every study time point, with multiple (e.g., five) replicate readings per site, averaged to obtain a single value per subject and visit. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; products are supplied in individual single-dose sa
Quantification of the change in facial skin hydration and transepidermal water loss (TEWL) from baseline to post-treatment visits using Corneometer® and Tewameter®. | Baseline (Day 0) and at approximately Day 28 (~4 weeks) and Day 56 (~8 weeks) of treatment.
  Sixty healthy women (35-65 years) with visible wrinkles in the crow's-feet area will take either a Collagen peptides supplement or a Competitor's collagen supplement once daily for 8 weeks. Skin hydration will be quantified with a Corneometer® CM 825 (Courage + Khazaka, Cologne, Germany), which measures changes in capacitance related to epidermal water content in the upper stratum corneum. TEWL will be assessed with a Tewameter® TM 300, based on an open-chamber method that calculates the water vapor gradient above the skin surface. Both parameters will be measured on the cheek of each volunteer at every study time point, with several replicate readings per subject and visit averaged to obtain a single value. Results will be expressed as absolute values and as percent change from baseline. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; products are supplied in individual single-dose sachets and stored according to the manufacturer's instructions.
Completion of a structured self-assessment questionnaire on perceived efficacy and skin appearance | Approximately Day 56 (~8 weeks) of treatment.
  Sixty healthy women (35-65 years) with visible wrinkles in the crow's-feet area will take either a Collagen peptides supplement or a Competitor's collagen supplement once daily for 8 weeks. Perceived efficacy will be evaluated using a structured self-assessment questionnaire completed by each participant after 56 days of treatment. Responses will be recorded on a 6-point Likert scale (1 = strongly disagree to 6 = strongly agree), with satisfaction for positive items defined as scores ≥4. For selected items, participants will provide binary yes/no answers. The questionnaire will capture subjective perceptions of changes in skin hydration, smoothness, firmness, wrinkle appearance, and overall skin quality. All procedures are conducted at Bionos Biotech S.L. facilities under a fixed schedule; products are supplied in individual single-dose sachets and stored according to the manufacturer's instructions.

CONTACTS AND LOCATIONS:
Overall Officials: Adela Serrano Gimeno, PhD, Principal Investigator — Bionos Biotech S.L. , LabAnalysis Life Science
Locations (1):
- Bionos Biotech S.L., LabAnalysis Life Science, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No